CLINICAL TRIAL: NCT00390078
Title: Single-Blind, Randomized, Controlled, Phase I/II Vaccination Study on Safety and Immunogenicity of a Recombinant MVA-HIV Polytope Vaccine (MVA-mBN32) in HIV-1 Infected Patients With CD4 Counts > 250/µl
Brief Title: Single-Blind, Controlled Safety and Immunogenicity Study of Recombinant MVA Virus to Treat HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Monika Fluer, Bavarian Nordic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIV-POL-002; NIAID Cont. No. N01-AI-40072
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: HIV Infections
Keywords: Vaccine; Safety; T-cell epitope; Acquired Immune Deficiency Syndrome Virus; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): 20 Subjects, 1x 10E8_TCID50 MVA-mBN32
  Interventions: Biological: MVA-mBN32
- 2 (Placebo Comparator): 10 Subjects 1x 10E8_TCID50 IMVAMUNE
  Interventions: Biological: IMVAMUNE

INTERVENTIONS:
Biological: MVA-mBN32 — 3 immunizations: 1x 10E8_TCID50 MVA-mBN32
  Arms: 1
Biological: IMVAMUNE — 3 immunizations: 1x 10E8_TCID50 IMVAMUNE
  Arms: 2

SUMMARY:
At the end of 2004 there were more than 40 million people infected Worldwide with HIV, with an estimated 16,000 new infections every day (UNAIDS, 2004). The HIV epidemic threatens whole societies particularly in Africa and Asia and rates of infections in the Western Countries have also increased over the last few years. However, despite more than 15 years of research, an effective vaccine against HIV and acquired immunodeficiency syndrome (AIDS) has still not been developed.

There is considerable evidence that cellular immune responses can effectively control HIV-1 replication during acute and chronic infections thereby possibly protecting individuals from infection and preventing the spread of HIV. To be truly effective in the general population, a vaccine must induce responses specific to immunologically conserved regions. The epitope-based vaccine MVA-mBN32 represent a very logical approach to this problem because its potential to elicit a polyfunctional immune response and to focus these responses to conserved epitopes.

In this study the safety, tolerability and immunogenicity of a recombinant MVA-BN® expressing CTL and HTL epitopes of HIV-1 (MVA-mBN32) vs. the vector control MVA-BN® in 30 HIV-infected subjects will be examined. This will include a full analysis of CD4+ T helper cells and CD8+ CTL responses to these epitopes, to establish the potential of such a homologous prime-boost vaccine approach to induce a broad cell-mediated response to different HIV antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18 to 50 years.
2. HIV-1 infection.
3. Stable on HAART with regard to immunologic and clinical parameters for at least 6 consecutive months prior to study entry.
4. Plasma HIV RNA level < 50 copies/ml for at least 6 months
5. Plasma HIV-1 RNA levels of < 50 copies/ml at study entry.
6. CD4 cells above 250/µl.
7. CD4 nadir > 200/µl.
8. HLA-A2, HLA-A3 or HLA-B7 positive.
9. Laboratory criteria (all of the following must be fulfilled):

   Adequate bone marrow reserve, Adequate renal function, Adequate hepatic function, Cardiac enzymes within normal range
10. For women, negative serum pregnancy test at screening and negative urine pregnancy test within 24 hours prior to each vaccination.
11. If the volunteer is female and of childbearing potential, she has used adequate contraceptive precautions for 30 days prior to the first vaccination and agrees to use an acceptable method of contraception, and not become pregnant for at least 56 days after the last vaccination.
12. Read, signed and dated informed consent document.

EXCLUSION CRITERIA:

1. Pregnancy or breast-feeding.
2. Uncontrolled serious infection
3. History of any serious medical condition, which in the opinion of the investigator, would compromise the safety of the subject.
4. History of or active autoimmune disease.
5. History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure.
6. History of chronic alcohol abuse (40g / day for at least 6 months) and/or intravenous drug abuse (within the past 6 month).
7. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
8. History of anaphylaxis or severe allergic reaction.
9. Acute disease (a moderate or severe illness with or without a fever) at the time of enrolment.
10. Any continuous therapy that may influence CD4 counts other than anti-retroviral therapy
11. Any vaccinations with live vaccines within a period starting 30 days prior to administration of the vaccine and ending 30 days after administration of the study vaccine. Any vaccinations with killed vaccines within a period starting 14 days prior to administration of the study vaccine and ending 14 days after administration of the study vaccine.
12. Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune-modifying drugs during a period starting from six months prior to administration of the vaccine and ending at study conclusion.
13. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at study conclusion.
14. Prior use of any HIV vaccine or vaccinia immunization within the last 5 years.
15. Use of any investigational or non-registered drug or vaccine.
16. History or clinical manifestation of clinically significant mental illness or severe haematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
17. ECG with clinical significance.
18. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
19. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to volunteers 20 years of age and older.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To compare the safety and reactogenicity of the recombinant MVA-mBN32 expressing functional HIV epitopes and MVA-BN® following repeated vaccination in HIV-1 infected patients | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Hain, PhD, Study Director — Bavarian Nordic
Locations (1):
- Charité, Campus Virchow-Klinikum, Berlin, Germany